CLINICAL TRIAL: NCT01926990
Title: Developing Non-Invasive Early Therapeutic Monitoring to Predict Treatment Efficacy in Renal Cell Carcinoma
Brief Title: Perfusion CT Monitoring to Predict Treatment Efficacy in Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Siemens Healthcare QT (Industry)
Responsible Party: Sponsor
Other Study IDs: RENAL0026; NCI-2013-01626 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Metastatic Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: perfusion computed tomography — Undergo perfusion CT
  Other Names: tomography, computed

SUMMARY:
This pilot clinical trial studies perfusion computed tomography (CT) in predicting response to treatment in patients with advanced kidney cancer. Comparing results of diagnostic procedures done before, during, and after targeted therapy may help doctors predict a patient's response to treatment and help plan the best treatment.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or biopsy-proven renal cell carcinoma
* Treatment planned with sunitinib, pazopanib, sorafenib, bevacizumab, axitinib, nivolumab alone or in combination with an investigational agent
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Serum creatinine greater than or equal to 1.7 mg/dL
* Severe allergy to contrast agent
* Any contraindication for undergoing a CT scan
* Pregnancy or unwillingness to use preventative measures if a woman of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with metastatic renal cell carcinoma prescribed a systemic targeted therapy medication
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2014-08; Primary Completion 2018-07-16 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Characterization of the relationship between Change in blood flow measured through perfusion CT techniques and Change in tumor size measured through non-investigational CT | 12 weeks (+/- 5 days) after start of standard systemic targeted therapy medication

SECONDARY OUTCOMES:
Characterization of the relationship between change in perfusion CT measurements (eg. Mean transit time) and change in tumor size measured by non-investigational CT | 12 weeks (+/- 5 days) after start of standard systemic targeted therapy medication
Relationship between change in blood flow and tumor response measured on ordinal scale | 12 weeks (+/- 5 days) after start of standard systemic targeted therapy medication
Relationship between change in blood flow at Day 8 and change in tumor size measured on continuous scale at Week 12 and tumor response measured on ordinal scale at Week 12 | 12 weeks (+/- 5 days) after start of standard systemic targeted therapy medication
Relationship between change in blood flow at Day 8 and at Week 12 and progression-free survival | 12 weeks after start of standard systemic targeted therapy medication
Relationship between change in blood flow at Day 8 and at Week 12 and time to nadir of tumor size | 12 weeks after start of standard systemic targeted therapy medication

CONTACTS AND LOCATIONS:
Overall Officials: Aya Kamaya, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University Cancer Institute, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No